CLINICAL TRIAL: NCT04290052
Title: Atrial Fibrillation on Holter Monitoring After Percutaneous Patent Foramen Ovale Closure : a Prospective Observational Study
Brief Title: Atrial Fibrillation After PFO Closure
Acronym: AFEPFO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0517
Record Dates: First submitted 2020-02-11; First posted 2020-02-28 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: Cryptogenic
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An increased risk of atrial fibrillation (AF) after patent foramen ovale (PFO) closure was observed in randomized trials but systematic screening of AF was not performed in these studies. Purpose: The objective of this study was to evaluate incidence of AF in patients who underwent percutaneous PFO closure with serial 24-hours ambulatory ECG (AECG) monitoring during 6 months follow-up. Primary endpoint was incidence of AF on ECG monitoring. Secondary endpoints were clinical outcomes (symptoms, hospitalization from cardiovascular causes, ischemic stroke, or bleeding) up to 6 month follow-up.

DETAILED DESCRIPTION:
This is a prospective, bicentric, observational cohort study which will be performed in University hospital center of Montpellier and Nîmes The study will include all consecutive patients, admitted for a percutaneous PFO closure after an ischemic stroke (IS) or a transient ischemic attack (TIA) of cryptogenic origin, or after the occurrence of a decompression illness during scuba diving. Patients eligible for the closure of a FOP in prevention of the recurrence of stroke or TIA of cryptogenic origin, was systematically evaluated for exclusion of supraventricular arrhythmia in accordance with international recommendations. This evaluation included a 12-lead ECG as well as an extended electrocardiographic monitoring lasting more than or equal to 24 hours (most frequently, performing a 72-hour ECG Holter). All patients previously has a transesophageal ultrasound (TEE) allowing to retain the diagnosis of PFO, to assess the presence or not of an atrial septum aneurysm (ASA) associated with PFO and to quantify the right to left shunt thanks to a contrast test potentiated by a Valsalva maneuver. Exclusion criteria included interatrial defect with left to right and others indications for PFO closure that cryptogenic stroke or decompression illness. Indication of PFO closure is always validated by a cardio neurological team.

The primary objective of the study was incidence of AF defined as an irregular rhythm without discernible P waves lasting at least 30 seconds on ECG monitoring during the 6-month follow-up. The secondary objectives were to evaluate the characteristics of the supra-ventricular arrhythmias (delay in onset, duration, recurrent nature), incidence of others arrhythmia, symptoms, and prognostic implications of AF (hospitalization , need of curative anticoagulation, need for cardioversion and occurrence of neurological accident documented by imagery (ischemic stroke or TIA). The investigators also evaluated risk factors for occurrence of arrhythmia.

A total of 100 patients included during 1 year is expected

ELIGIBILITY:
Inclusion Criteria:

* Men or women over the age of 18 to 60
* Benefiting from the closure of the FOP percutaneously after a cryptogenic ischemic stroke or a TIA (indication validated during a multidisciplinary meeting with neurologists and cardiologists)

Exclusion Criteria:

* Inability to perform a 24h ECG Holter
* Pregnant or lactating women
* Vulnerable people

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient at least 18 years old, benefiting from percutaneous closure of the FOP after a cryptogenic stroke (indication validated during a multidisciplinary meeting with neurologists and cardiologists)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
occurrence of sustained supra-ventricular arrhythmia | the 24-hour post-intervention
  occurrence of sustained supra-ventricular arrhythmia (AF, atrial flutter) during the analysis the 24-hour Holter ECG performed post-intervention
occurrence of sustained supra-ventricular arrhythmia | at 1 month
  occurrence of sustained supra-ventricular arrhythmia (AF, atrial flutter) during the analysis at 1 month (Holter ECG)
occurrence of sustained supra-ventricular arrhythmia | at 6 month
  occurrence of sustained supra-ventricular arrhythmia (AF, atrial flutter) during the analysis at 6 month (Holter ECG)
occurrence of sustained supra-ventricular arrhythmia | at 12 month
  occurrence of sustained supra-ventricular arrhythmia (AF, atrial flutter) during the analysis at 12 month (Holter ECG)

SECONDARY OUTCOMES:
characteristics of these detected arrhythmias | 24 hours post-intervention to 12 months
  characteristics of these detected arrhythmias : time to onset
characteristics of these detected arrhythmias | 24 hours post-intervention to 12 months
  characteristics of these detected arrhythmias : duration
characteristics of these detected arrhythmias | 24 hours post-intervention to 12 months
  characteristics of these detected arrhythmias : recurrence
symptoms related to the arrhythmia episode | 24 hours post-intervention to 12 months
  symptoms related to the arrhythmia episode
hospitalization related to arrhythmia | 24 hours post-intervention to 12 months
  hospitalization related to arrhythmia
occurrence of a neurological accident. | 24 hours post-intervention to 12 months
  occurrence of a neurological accident.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC